CLINICAL TRIAL: NCT00001574
Title: A Pilot Study of 1H-Nuclear Magnetic Resonance Spectroscopic Imaging in Pediatric Patients With Primary and Metastatic Brain Tumors
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970093; 97-C-0093; NCT00019292 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05-06

CONDITIONS: Brain Neoplasm; Brain Cancer; Brain Tumor, Primary
Keywords: Metabolites; Proton Nuclear Magnetic Resonance Spectroscopic Imaging; Scans
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Brain tumors represent the most common solid tumor of childhood. Treatment generally entails surgery and radiation, but local recurrence is frequent. Chemotherapy is often used in an adjuvant setting, to delay radiation therapy or for resistant disease. Children with brain tumors are generally followed by imaging studies, such as CT or MRI. Difficulty arises in trying to distinguish tumor regrowth from treatment related edema, necrosis or radiation injury. Proton Nuclear Magnetic Resonance Spectroscopic (NMRS) Imaging is a non-invasive method of detecting and measuring cellular metabolites in vivo. NMRS imaging complements routine MRI by giving chemical information in conjunction with spatial information obtained by MRI.

This study will be conducted to determine NMRS imaging patterns before, during and after chemotherapy in pediatric patients with primary or metastatic brain tumors in an attempt to identify and characterize specific patterns of metabolites related to tumor regrowth, tumor response to therapy, edema or necrosis.

DETAILED DESCRIPTION:
Background:

* Brain tumors represent the most common solid tumor of childhood. Treatment generally includes surgery and radiation, but recurrences are frequent, particularly for high-grade lesions.
* Chemotherapy is often used in an adjuvant setting, to delay radiation therapy or for resistant disease.
* Children with brain tumors are generally followed by imaging studies, such as CT or MRI.
* Difficulty arises in trying to distinguish tumor regrowth from treatment related edema, necrosis or radiation injury.
* Proton Nuclear Magnetic Resonance Spectroscopic (NMRS) Imaging is a non-invasive method of detecting and measuring cellular metabolites in vivo.

Objective:

* To determine NMRS imaging patterns before, during and after chemotherapy in pediatric patients with primary or metastatic brain tumors
* To identify and characterize specific patterns of metabolites related to tumor regrowth, tumor response to therapy, edema or necrosis.

Eligibility:

* Age less than or equal to 21 years.
* Patients entered on this trial will also be entered on one of the Branch s primary brain tumor treatment trials.
* Histologically confirmed primary or metastatic brain tumor. Patients with a brainstem glioma or optic pathway gliomas are not required to have a histologic diagnosis.
* Measurable or evaluable tumor at the time of study entry.

Design:

* This is intended to be a pilot study to define metabolite patterns associated with tumor growth, tumor edema and tumor necrosis as seen on standard MRI; and determine the feasibility of using metabolite patterns to predict response to therapy in pediatric patients with brain tumors.
* Contalateral spectroscopic analysis of normal appearing brain will also be performed when feasible.
* Analysis of results will be stratified according to type of tumor, and prior history of radiation therapy or surgery.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age less than or equal to 21 years.

Patients entered on this trial will also be entered on one of the Pediatric Oncology Branch's primary treatment trials (e.g., phenylacetate, phenylbutyrate, SU-101) or on the Natural History or Standard Therapy protocols. The patient's management will be determined by the primary treatment protocol.

Histology confirmed primary or metastatic brain tumor. Patients with a brainstem glioma are not required to have previously had a histologic diagnosis.

Measurable or evaluable tumor at the time of study entry.

Durable Power of Attorney (DPA): A DPA is required of all patients 18 - 21 years of age.

All patients or their legal guardians (if the patient is less than 18 years of age) must sign a document of informed consent indicating their awareness of the investigational nature and the risks of this study. When appropriate the minor patient will give verbal assent.

EXCLUSION CRITERIA:

Pregnant women.

Any patient who is unable (either because of physical or psychological factors) to undergo imaging studies and who is not an anesthesia candidate.

Any patient with a metallic implant, including cardiac pacemakers, neural pacemakers, shrapnel, cochlear implants or ferrous surgical clips.

Any patient with a history of a severe reaction to Gadolinium or other contrast agents.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 1997-03-14; Study Completion 2019-05-06

PRIMARY OUTCOMES:
To define specific patterns of metabolises using long-echo time multislice proton nuclear magnetic resonance spectroscopic imaging in pediatric patients with brain tumors. | at time of disease evaluation
  in vivo measurements of tissue metabolites (NAA, Cho,Cr, Lac) and what they reflect

SECONDARY OUTCOMES:
Distinguish spectroscopic patterns associated with tumor progression, necrosis and edema | at time of disease evaluation
  measurements and differences of signal intensity of peaks obtained for tissue metabolites (NAA, Cho, Cr, Lac)
Determine if early metabolic changes are predictive of response | at time of disease evaluation
  Contalateral spectroscopic analysis results, stratified according to type of tumor, history of radiation therapy or surgery

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Castillo M, Kwock L, Mukherji SK. Clinical applications of proton MR spectroscopy. AJNR Am J Neuroradiol. 1996 Jan;17(1):1-15. No abstract available. PMID 8770242
- [Background] Sutton LN, Wang Z, Gusnard D, Lange B, Perilongo G, Bogdan AR, Detre JA, Rorke L, Zimmerman RA. Proton magnetic resonance spectroscopy of pediatric brain tumors. Neurosurgery. 1992 Aug;31(2):195-202. doi: 10.1227/00006123-199208000-00004. PMID 1513425
- [Background] Duyn JH, Gillen J, Sobering G, van Zijl PC, Moonen CT. Multisection proton MR spectroscopic imaging of the brain. Radiology. 1993 Jul;188(1):277-82. doi: 10.1148/radiology.188.1.8511313.